CLINICAL TRIAL: NCT05615324
Title: The Randomized Clinical Trial SAFIR FAMILY TALK: a Short Family-based Early Intervention vs. Service as Usual for Children of Parents With Mental Illness in the Capital Region of Denmark
Brief Title: SAFIR Family Talk - Investigating the Effect of The Family Talk Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: TrygFonden, Denmark (Industry); Sektion for Tværsektoriel forskning - Region Hovedstaden (Unknown)
Responsible Party: Principal Investigator, Anne Ranning, Assistant Professor, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 127849
Record Dates: First submitted 2022-10-26; First posted 2022-11-14 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Mental Disorder; Family; Child; Parenting; Resilience; Prevention
Keywords: Parental mental illness; COPMI; Intervention; Family Talk; Mental Illness; Beardslee
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: SAFIR Family Talk is i randomized controlled trial carried out in the capital region of Denmark. The trial examines the Family Talk intervention, developed by William Beardslee, as opposed to service as usual (SAU) in out patient clinics in the public health sector in the capital region of denmark. All participating families will be assessed at baseline, 4 months follow-up and 12 months follow-up.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The research assistants and ph.d.-students in charge of the assessment are blinded in regards to which treatment the families have received. All outcome scores are set in consensus with the other outcome assessors. In case of unblinding, it is the team setting the score, not the assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Talk (Experimental): families will receive a manualized, family-based intervention Family Talk of approximately 8 sessions with a trained, Family Talk interventionist.
  Interventions: Behavioral: Family Talk Preventive Intervention
- Service as usual (No Intervention): Families in this arm will not receive any intervention from the research team but they may receive other services. It is likely that many will receive two sessions of talk intervention concerning parental mental health and child well-being from professionals in the mental health sector where the parent is treated.

INTERVENTIONS:
Behavioral: Family Talk Preventive Intervention — This is a clinician facilitated, psychoeducational preventive intervention that includes on average 8 sessions designed to improve family communication and understanding of parental mental illness, improve interpersonal relationships, and promote child resilience and utilization of social support. An important tool throughout the intervention is the logbook which the clinician uses for taking notes with each family. The logbook prescribes the planned topics to be covered in each session and the contents of the sessions are noted in the logbook by the clinicians.
  Other Names: Beardslee's Family Intervention
  Arms: Family Talk

SUMMARY:
The goal of this clinical trial is to test the effect of the Family Talk Preventive Intervention compared to service as usual for families where a parent has mental illness. Participants are the parent with a mental illness receiving treatment from a secondary mental health service within the last two years from inclusion, their youngest child aged 7-17 years and the other parent of this child. The main questions it aims to answer are:

Is Family Talk superior to service as usual regarding improving?

* The child's level of functioning
* The parent's sense of competence
* Family functioning Participants will undergo interviews and fill out questionnaires. Half will be randomized to Family Talk and receive a manualized, family-based intervention of approximately 8 conversations with a trained, Family Talk interventionist. The other half will be randomized to service as usual which is normally two conversations with a professional in the mental health sector. The researchers will compare the two groups on child's level of functioning, parental sense of competence and family functioning.

DETAILED DESCRIPTION:
Children of parents with mental illness are at increased risk for mental illness themselves and therefore interventions aimed at mitigating this risk are important. The Family Talk Preventive Intervention was developed by William Beardslee in the 1980's for families with parental depression but has been widely used to treat families with other mental health conditions as well. Nevertheless, only few high-quality clinical trials exist, and the results are inconclusive.

The objective of this clinical trial is to test the effect of Family Talk Preventive Intervention compared to service as usual for families where a parent has mental illness and receiving treatment from a secondary mental health service within the last two years from inclusion. Participants are the parent with a mental illness, their youngest child aged 7-17 years and the other parent of this child. The hypothesis is that Family Talk will be superior to service as usual in improving the child's level of functioning, the parent's sense of competence and family functioning at 4 moths follow-up.

Participants will undergo interviews and fill out questionnaires at baseline, four- and twelve months follow-up assessments. Half of the families will be randomized to Family Talk and receive a manualized, family-based intervention of approximately 8 conversations with a trained, Family Talk interventionist. The other half will be randomized to service as usual which is normally two conversations with a professional in the mental health sector. The researchers will compare the two groups on child's level of functioning, parental sense of competence and family functioning and other measures including child's quality of life, communication in the family and parental personal recovery.

ELIGIBILITY:
Inclusion Criteria:

* At least one parent must have been in contact with the secondary health care system due to a mental health condition within the last two years before inclusion.
* The parent should have at least one child aged 7-17 years at the time of inclusion.
* The other parent of this child may or may not have a mental health condition.

Exclusion Criteria:

- Not speaking Danish or English.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Children's Global Assessment Scale (CGAS) | Assessment at baseline, 4 months and 12 months after baseline.
  A clinician rated measurement to asses general functioning in children. Information is obtained from both the child and the parents. Scale from 1-100. High score indicates better the functioning.
Change in Family Assessment Device (FAD) (Parent-rated) | Assessment at baseline, 4 months and 12 months after baseline.
  A 60 item parent report questionnaire assessing each individual's perception of his or her family functioning. The FAD is based on a comprehensive sociological theory about different functions of a family. Scale from 1-4. Low score represents better outcome.
Change in Parenting Sense of Competency (PSOC) | Assessment at baseline, 4 months and 12 months after baseline.
  A 16 item parent report questionnaire assessing overall parenting sense of competence. Each item rated on a 6-point Likert scale. Total scale from 16-96. A higher score indicates a higher parenting sense of competency.

SECONDARY OUTCOMES:
Change in Beck's Youth Inventories (BYI-II) | Assessment at baseline, 4 months and 12 months after baseline.
  A 99 item self report measure consisting of 5 subscales to assess symptoms of Depression, Anxiety, Anger, Disruptive behaviour and Self-concept in children. Higher scores are associated with negative affect.
Change in Parent-Child Communication (Child-rated) | Assessment at baseline, 4 months and 12 months after baseline.
  Questionnaire assessing communication between the child and the mentally ill parent. A 10 item questionnaire for children ages 8-12 and a 19 item questionnaire for children ages 13-17. Each item rated on a 6-point Likert scale. A higher score indicates better communication.
Change in Response to parents' mood | Assessment at baseline, 4 months and 12 months after baseline.
  A 4-questions multiple-choice questionnaire administered to the child assessing the child's reaction to the parents' mood.
Change in parental recovery (Brief INSPIRE-O) | Assessment at baseline, 4 months and 12 months after baseline.
  A 5 item self-report questionnaire completed by the parents assessing personal recovery. Each item rated on a score from 0-100. A higher score indicates better recovery.

OTHER OUTCOMES:
Change in Child-rated Strengths and Difficulties Questionnaire (SDQ) | Assessment at baseline, 4 months and 12 months after baseline.
  A 25 item self-report questionnaire assessing developmental, behavioural and emotional problems completed by children aged 11-17. Items are rated on a three-point Likert scale (0= not true, 1= somewhat true, 2= certainly true).
Change in Parent-rated Strengths and Difficulties Questionnaire (SDQ) | Assessment at baseline, 4 months and 12 months after baseline.
  A 25 item questionnaire assessing developmental, behavioural and emotional problems in children completed by the Primary-Caregiver as a respondent. Items are rated on a three-point Likert scale (0= not true, 1= somewhat true, 2= certainly true).
Change in children's Quality of Life (Kidsscreen-27) | Assessment at baseline, 4 months and 12 months after baseline.
  A 27 item self-report questionnaire assessing health related Quality of Life completed by the child. Each item is rated on a 5-point Likert scale. A higher score indicates a better quality of life.
Change in Child and Youth Resilience Measurement (CYRM) | Assessment at baseline, 4 months and 12 months after baseline.
  A 12 item self-report questionnaire assessing resiliency in children across a number of areas including personal skills, peer support, social skills, physical and psychological caregiving, educational and cultural. Items are rated on a 3- or 5-point Likert scale. Higher scores indicating greater resiliency.
Change in Guilt and Shame Questionnaire (GSQ-AMPI) | Assessment at baseline, 4 months and 12 months after baseline.
  A 10 item self-report questionnaire completed by the child assessing feelings of guilt and shame in children of parents with mental illness. Items are rated on a 5-point Likert scale. Higher scores indicate higher feelings of guilt or shame.
Change in Personal and Social Performance (PSP) | Assessment at baseline, 4 months and 12 months after baseline.
  An interviewer-rated scale assessing the Parents personal and social functioning over four domains such as social activities, relationships, self-care and aggressive behavior. The PSP provides a global score on a scale from 1-100, with lower scores indicating lower social functioning.
Change in Global Assessment of Functioning (GAF-S) | Assessment at baseline, 4 months and 12 months after baseline.
  An interviewer-rated scale assessing the Parents Level of Psychiatric Symptoms. GAF-S provides a score from 1-100, with higher scores indicating better outcome.
Change in Parent-Child Communication (Parent-rated) | Assessment at baseline, 4 months and 12 months after baseline.
  A 19 or 20 item questionnaire completed by the parents assessing communication between the parent and the child. Each item rated on a 5-point Likert scale. A higher score indicates better communication.
Family Talk Evaluation Questionnaire (Child-rated) | Assessment at 4 months after baseline where the families have completed the SAFIR Family Talk Intervention.
  A 9 item self report questionnaire only administered to children from the SAFIR Family Talk Intervention group to assess their experience of the intervention.
Family Talk Evaluation Questionnaire (Parent-rated) | Assessment at 4 months after baseline where the families have completed the SAFIR Family Talk Intervention.
  A 68 item self report questionnaire only administered to parents from the SAFIR Family Talk Intervention group. The questionnaire assess the parents experience of the intervention across a number of areas including the therapeutic alliance, client satisfaction and negative effects of the intervention. Each item rated on a 5-point Likert scale. A higher score indicates better outcome.
Working Alliance Inventory (WAI) | Assessment at 4 months after baseline where the families have completed the SAFIR Family Talk Intervention.
  A 12 item questionnaire only administered to parents from the SAFIR Family Talk Intervention group to assess key aspects of the therapeutic alliance. Each item are rated on a 7-point Likert scale. Scale from 12-84. A higher score indicates better outcome.
Client Satisfaction Questionnaire (CSQ-8) | Assessment at 4 months after baseline where the families have completed the SAFIR Family Talk Intervention.
  A 8 item questionnaire only administered to parents from the SAFIR Family Talk Intervention group to assess the parents' experiences with different objectives in the intervention. Each item is rated on a 4-point Likert scale. Scale from 8-32. A higher score indicates greater satisfaction.
Negative effects of the intervention assessed with the Negative Effects Questionnaire (NeQ) | Assessment at 4 months after baseline where the families have completed the SAFIR Family Talk Intervention.
  A 21 item questionnaire only administered to parents from the SAFIR Family Talk Intervention group to investigate negative effects of the intervention. Each item is answered by "yes" or "no", where "yes" indicates better outcome.
Change in child's number of days absent from school | Assessment at baseline, 4 months and 12 months after baseline.
  Number of days the child was absent from school within the last 3 months. Low number represent better outcome. Information will be obtained from registry and parents' report.
Change in The McMaster Family Assessment Device (FAD) (Children self-report) | Assessment at baseline, 4 months and 12 months after baseline.
  A 60 item self-report only administered to children ages 12-17 assessing family functioning. Scale from 1-4. Low score represents better outcome.
Change in Children of Parents with Mental Illness Questionnaire (COPMI-Q) | Assessment at baseline, 4 months and 12 months after baseline.
  A 16 item questionnaire assessing the child's concerns regarding the mentally ill parent and thoughts on mental illness. Each item is rated on a 3-point Likert scale. A higher score indicates a more positive outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Ranning, PhD, Principal Investigator — Mental Health Services in the Capital Region of Denmark
Locations (1):
- Mental Health Services in the Capital Region, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nielsen SS, Mikkelsen LJ, Quaade N, Gladstone TRG, Beardslee WR, Bonnemose K, Rosenberg NK, Hjorthoj C, Thorup AAE, Nordentoft M, Ranning A. A study protocol for the randomized controlled trial SAFIR FAMILY TALK: a selective primary preventive intervention vs. service as usual for children of parents with mental illness. Trials. 2023 Apr 22;24(1):291. doi: 10.1186/s13063-023-07256-6. PMID 37087437

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-07-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT05615324/SAP_001.pdf